CLINICAL TRIAL: NCT05038020
Title: A Double-Masked, Placebo-Controlled Study to Evaluate the Efficacy of Oral AKST4290 in Participants With Moderately Severe to Severe Diabetic Retinopathy (CAPRI)
Brief Title: A Study to Evaluate the Efficacy of Oral AKST4290 in Participants With Moderately Severe to Severe Diabetic Retinopathy (CAPRI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to safety findings in other AKST4290 studies
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKST4290-231
Record Dates: First submitted 2021-07-29; First posted 2021-09-08 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Retinopathy
Keywords: CCR3 inhibition; Diabetic Retinopathy; Oral Treatment
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AKST4290 (Experimental): Subjects will receive AKST4290, 400mg twice daily, for 24 weeks
  Interventions: Drug: AKST4290
- Placebo (Placebo Comparator): Subjects will receive matching Placebo, twice daily, for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AKST4290 — Oral AKST4290
  Arms: AKST4290
Drug: Placebo — Oral Placebo
  Arms: Placebo

SUMMARY:
A Double-Masked, Placebo-Controlled Study to Evaluate the Efficacy of Oral AKST4290 in Participants with Moderately Severe to Severe Diabetic Retinopathy (CAPRI).

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy of AKST4290 administered at a total daily dose (TDD) of 800 mg daily (400 mg twice daily [b.i.d.]) compared with placebo over a 24-week dosing period in participants with moderately severe non-proliferative diabetic retinopathy (NPDR) to severe NPDR.

Participants will be enrolled and allocated to 1 of 2 treatment arms in a 2:1 randomization scheme (AKST4290: placebo). Participants will receive treatment for a total of 24 weeks with either AKST4290 800 mg daily (400 mg b.i.d.) in Arm 1 or placebo (matching tablets) in Arm 2

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Type 1 or type 2 DM.
3. BCVA ETDRS visual acuity letter score≥ 69 letters at Screening.
4. Moderately severe NPDR (DRSS Level 47) to severe NPDR (DRSS Level 53).

Exclusion Criteria:

1. Evidence of neovascularization (NV) (including active iris or angle NV) requiring treatment, per investigator discretion.
2. PRP or grid laser within 1000 microns of the foveal center.
3. Center-InvolvedI-Diabetic Macular Edema (CI-DME) on clinical examination (CI is defined as DME within 1,000 microns of the foveal center).
4. Prior Intraocular of periocular steroid Injection
5. Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to enrollment and assignment to a randomized treatment.
6. History of vitreoretinal surgery.
7. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
8. History of DME or DR treatment with laser or intraocular injections of medication.
9. Medical history or condition that, in the opinion of the investigator would preclude participation in the study.
10. Clinically relevant abnormal laboratory value at Screening, including hematology, blood chemistry, or urinalysis (laboratory testing may be repeated once during the Screening phase).
11. Malignancy for which the participant has undergone resection, radiation, or chemotherapy within the past 5 years (treated basal cell carcinoma or fully cured squamous cell carcinoma are allowed).
12. Concurrent participation in another interventional clinical trial; prior clinical trial participants must have been off study agents for at least 30 days for small molecules, 4 months for disease modifying therapies, and 1 year for vaccine or immunotherapy trials prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (17):
- United States (17):
  - Site 132, Phoenix, Arizona
  - Site 136, Phoenix, Arizona
  - Site 123, Glendale, California
  - Site 121, Huntington Beach, California
  - Site 116, Clearwater, Florida
  - Site 117, Sarasota, Florida
  - Site 118, Winter Haven, Florida
  - Site 120, Oak Forest, Illinois
  - Site 133, Beaufort, South Carolina
  - Site 127, Ladson, South Carolina
  - Site 122, Arlington, Texas
  - Site 130, Bellaire, Texas
  - Site 126, Harlingen, Texas
  - Site 134, Houston, Texas
  - Site 129, Katy, Texas
  - Site 128, San Antonio, Texas
  - Site 125, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early by the Sponsor. At the time of discontinuation, three participants were enrolled and none completed the study.
Period: Overall Study
Arm/Group | AKST4290 | Placebo
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Early Termination | 3 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor. Only 3 participants were enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | AKST4290 | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Diabetes Mellitus Type

OUTCOME MEASURES:

1. Primary Outcome: To Investigate the Efficacy of AKST4290 Assessed by the Improvement in the DRSS Score From Baseline.
Description: The Diabetic Retinopathy Severity Scale (DRSS) divides DR into 13 levels ranging from the absence of retinopathy to severe retinopathy and is used to describe overall DR severity as well as the change in severity over time. Higher scores indicate more severe DR.
  To be eligible for the study, participants needed to have moderately severe non-proliferative DR (NPDR) (DRSS Level 47) to severe NPDR (DRSS Level 53) in one eye, and at least mild NPDR (DRSS Level 35) to mild proliferative DR (PDR) (DRSS Level 61) in the other eye at baseline.
  The DRSS score is derived from fundus photography (FP) and fluorescein angiography (FA) findings.
  The primary efficacy endpoint is the proportion of participants with a ≥ 3-step improvement from baseline on the DRSS score as compared with Week 24.
Time Frame: Baseline to Week 24
Population: as for baseline characteristics
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Investigate Additional Measures of Efficacy of AKST4290 Assessed by the Improvement in the DRSS Score From Baseline.
Description: The Diabetic Retinopathy Severity Scale (DRSS) divides DR into 13 levels ranging from the absence of retinopathy to severe retinopathy and is used to describe overall DR severity as well as the change in severity over time. Higher scores indicate more severe DR.
  The DRSS score is derived from fundus photography (FP) and fluorescein angiography (FA) findings.
  The secondary efficacy endpoint is the proportion of participants with a ≥ 2-step improvement from baseline on the DRSS score as compared with Week 24.
Time Frame: Baseline to Week 24 or 28
Population: as for baseline characteristics
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Assess the Proportion of Participants Progressing to (or Worsening of) Center-involved Diabetic Macular Edema (CI-DME), Proliferative Diabetic Retinopathy (PDR), and/or Anterior-segment Neovascularization (ASNV).
Description: The secondary efficacy endpoint is the proportion of participants progressing to the following vision-threatening complications that require treatment: CI-DME, PDR, and/or ASNV as assessed by spectral domain optical coherence tomography (SD-OCT), fundus photography (FP), and fluorescein angiography (FA), as appropriate. The central reading center must confirm progression to CI-DME and PDR before treatment is initiated; progression to ASNV, and subsequent treatment, does not require photo documentation.
Time Frame: Baseline to Week 28
Population: as for baseline characteristics
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Assess the Time to Event of CI-DME, PDR, and/or ASNV Requiring Treatment.
Description: The secondary efficacy endpoint is the time to the following vision-threatening event(s) that require treatment: CI-DME, PDR, and/or ASNV
Time Frame: Baseline to Week 28
Population: as for baseline characteristics
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Assess the Overall Safety of AKST429
Description: Safety was assessed based on the number of participants who reported adverse events of mild, moderate or severe intensities.
Time Frame: Baseline to Week 28
Population: The study was terminated early by the Sponsor. At the time of discontinuation, three participants were enrolled, and all participants were allocated to randomized treatment with AKST4290.
Measure: Count of Participants; unit: Participants
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 3 | 0
Participants
  AE Intensity - Mild | 1 | 0
  AE Intensity - Moderate | 2 | 0
  AE Intensity - Severe | 0 | 0

6. Secondary Outcome: To Assess the Effect of AKST4290 on Diabetic Kidney Disease
Description: The secondary efficacy endpoint is the effect of AKST4290 on diabetic kidney disease as assessed by changes in clinical laboratory values over time (eg, estimated glomerular filtration rate [eGFR], urine albumin to creatinine ratio [UACR]).
Time Frame: Baseline to Week 28
Population: as for baseline characteristics
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Evaluate the Changes From Baseline in the Workplace Productivity and Activity Impairment General Health (WPAI-GH) Questionnaire.
Description: The WPAI-GH V2.0 is a 6-question survey used to assess the effects of a participant's health problems (i.e., physical or emotional problems or symptoms) on their ability to work and perform regular activities during the past seven days. The WPAI-GH questions will be analyzed as impairment percentages, in which higher percentages indicate greater impairment and less productivity.
  The following parameters will be calculated (multiply scores by 100 to express in percentages):
  * Percent of work time missed due to health: Q2 divided by (Q2 plus Q4)
  * Percent of impairment while working due to health: Q5 divided by 10
  * Percent of overall work impairment due to health: Q2 divided by (Q2 plus Q4) plus [(1 - (Q2 divided by (Q2 plus Q4 ))) multiplied by (Q5 divided by 10)]
  * Percent of activity impairment due to health: Q6 divided by 10
Time Frame: Baseline to Week 24
Population: as for baseline characteristics
Arm/Group | AKST4290 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The planned timeframe for adverse event (AE) collection was from the first dose of the study drug until the post-treatment follow-up period (baseline to Week 28). However, the study was terminated early by the sponsor. At the time of termination, 3 participants were enrolled and none completed the study. Enrolled subjects had a safety visit at 30 and 60 days following study drug discontinuation.
Description: Three participants were enrolled and none completed the study. All participants were allocated to randomized treatment with AKST4290, and no participants received placebo.
Arm/Group | AKST4290 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 2/3 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AKST4290 (N=3) | Placebo (N=0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Worsening of Diabetes
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) — Elevated APTT on labs

LIMITATIONS AND CAVEATS:
This study was terminated by the Sponsor. Only 3 participants were enrolled in this study. Based on low enrollment number, no data is reported in order to protect and maintain participant privacy/confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT05038020/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT05038020/SAP_001.pdf